CLINICAL TRIAL: NCT01099020
Title: Temporal Pattern of Circulating DNA for Patients Receiving Total Body Irradiation
Brief Title: Temporal Pattern of Circulating DNA for Patients Receiving Irradiation
Status: Terminated | Type: Observational
Why Stopped: Funding for project was withdrawn
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michael Milano, MD,PhD, Principal investigator, University of Rochester
Other Study IDs: ULAB10008
Record Dates: First submitted 2010-04-02; First posted 2010-04-06 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Radiation
Keywords: Subjects receiving large volumes of Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the research study is to test a measurement tool that will determine the radiation dose people receive when they have been accidentally exposed to radiation. This test will be done using a small amount of blood and known dose of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be scheduled to undergo Total Body Irradiation (TBI) as part of a conditioning regime for a Bone Marrow Transplant. OR, Be scheduled to undergo Radiation Therapy treatment for a malignancy or other disease and have a radiation treatment field that contains at least 2 liters of tissue receiving at least 2 Gy radiation dose over the first 5 days of treatment.
* Patient must be willing to have blood draws as defined below.
* Patient must provide study-specific informed consent prior to study entry.
* Hemoglobin≥8.
* Age ≥ 18, but not older than age 60.

Exclusion Criteria:

* Patients not meeting the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving large volume of radiation for the treatment of their cancer
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States